CLINICAL TRIAL: NCT03962621
Title: A Randomized Controlled Trial of the Efficacy of a Non-ablative Erbium:YAG 2940nm in Combination With 1064nm Laser on Facial Rejuvenation
Brief Title: A Study of the Efficacy of Erbium:YAG 2940nm in Combination With 1064nm Laser on Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xjpfW (Other)
Collaborators: Air Force General Hospital of the PLA (Other Government); First Hospital of China Medical University (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, xjpfW, Head of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: XijingH-PF-20161117
Record Dates: First submitted 2019-05-10; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Facial Rejuvenation
Keywords: Facial rejuvenation, Erbium: YAG Laser, 1064 nm laser, skin aging
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2940 nm group (Active Comparator): Subjects were randomly assigned into two groups (n=10 per group) based on a treated with a Fotona 4D 2940 nm laser alone, the other side of face was treated with a Fotona 4D 2940 nm in combination with 1064 nm laser. The patients received three treatment sessions with monthly intervals between each session.
  Interventions: Radiation: Fotona 4D 2940 nm laser
- 1064 nm group (Active Comparator): Subjects were randomly assigned into two groups (n=10 per group) based on a treated with a Fotona 4D 1064 nm laser alone, the other side of face was treated with a Fotona 4D 2940 nm in combination with 1064 nm laser. The patients received three treatment sessions with monthly intervals between each session.
  Interventions: Radiation: Fotona 4D 1064 nm laser
- Combined treatment group (Experimental): Subjects were randomly assigned into two groups (n=10 per group) based on a treated with a Fotona 4D 2940 nm or 1064 nm laser (Fotona, Slovenia, EU) alone, the other side of face was treated with a Fotona 4D 2940 nm in combination with 1064 nm laser. The patients received three treatment sessions with monthly intervals between each session.
  Interventions: Radiation: Fotona 4D 1064 nm laser; Radiation: Fotona 4D 2940 nm laser

INTERVENTIONS:
Radiation: Fotona 4D 1064 nm laser — The 1064 nm laser can penetrate deep into the skin to explode pigment particles, destroy blood vessels and heat the dermal collagen by targeting melanin and haemoglobin.(1) Frac3®: 30-35 J/cm2, 1.6 ms pulse width, 4mm spot size, unilaterally accumulated 2000 shots; and (2) PIANO®: 160 J/cm2, 5s pulse width, spot size 9mm, unilaterally accumulated 20000 shots, to increase and maintain facial skin temperature to 39-40oC.
  Arms: 1064 nm group; Combined treatment group
Radiation: Fotona 4D 2940 nm laser — Er:YAG 2940nm have been considered as a good treatment of facial aging, especially in wrinkles.(1) Smooth®: 9-10 J/cm2, 7mm spot size, which is sequentially delivered to upper and lower labial mucosa and buccal mucosa to unilaterally accumulate 5000 shots; (2) SupErficial™: 0.5-1.0 J/cm2, 7mm spot size, a single pass
  Arms: 2940 nm group; Combined treatment group

SUMMARY:
1. Facial aging is a progressive, multifactor-induced and multidimensional process which is naturally irreversible. The prominent clinical features of skin aging include loss of volume, pigmentation irregularity, low light reflectance, static and dynamic wrinkles, etc.
2. The development of superpulsed CO2 and Erbium: YAG 2940 nm resurfacing lasers was considered as the "gold standard" for the treatment of facial aging [8,9]. However, many drawbacks including intraoperative pain, post procedural erythema, edema, high risk of changes of pigmentation and long downtime have drawn concerns to patients and practitioners. Therefore, the facial rejuvenation therapies based on combined modalities to target various factors simutaneously have raised more and more interests.
3. The Fotona 4D laser platform incorporates the long pulsed 1064 nm and 2940 nm lasers, which provides versatile modalities to target various skin aging problems simultaneously. The 1064 nm laser can penetrate deep into the skin to explode pigment particles, destroy blood vessels and heat the dermal collagen by targeting melanin and haemoglobin. The 2940 nm Er:YAG laser in Fotona 4D system integrates a non-ablative Smooth® mode and cold peel SupErficial™ mode. the half-face treated by a 2940 nm laser alone showed a significant improvement on indexes of skin wrinkles, texture, pores and elasticity as compared to the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients ranged in age from 35 to 60 years old.
* Patients had Dover scale between 2-4
* Fitzpatrick wrinkles scale between 1-3
* medium to very severe nasolabial fold depression with morphological scores of 2 - 3 points.

Exclusion Criteria:

* pregnancy,
* liver or kidney functional abnormality,
* skin ulceration
* skin cancer
* coagulation disorders
* patients on drugs of photosensitizing or anticoagulation agents
* systemic diseases such as cardiovascular disease, epilepsy, diabetes.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Visia CR imaging system | change from week0 to week24
  With fast capture times and lighting modes designed to enhance the visualization of skin features, VISIA®-CR (Canfield Scientific, Inc. USA) is the standard in repeatable clinical imaging. Visia CR imaging system can be used to assess the skin wrinkles, and elasticity

SECONDARY OUTCOMES:
Multiprobe skin testing system | change from week0 to week24
  Multiprobe skin testing system (CK, Germany) is used to detect skin elasticity

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital

IPD SHARING:
Plan to Share IPD: No